CLINICAL TRIAL: NCT01170351
Title: Comparing Efficacy and Tolerability of Cyclosporine-A vs. Prednisolone for Induction of Remission in Auto-immune Hepatitis
Brief Title: Cyclosporine-A Versus Prednisolone for Induction of Remission in Auto-immune Hepatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Siavosh Nasseri-Moghadam, MD, MPH, AGAF, Associate Professor of Medicine, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DDRC-301174
Record Dates: First submitted 2010-07-24; First posted 2010-07-27 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Autoimmune Hepatitis
Keywords: autoimmune hepatitis; corticosteroids; cysclosporine-A; treatment; treatment-naive; induction of remossion; efficacy; tolerability
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group-A (Active Comparator): Treatment-naive AIH patients consenting to participate
  Interventions: Drug: Cyclosporine-A
- Group-B (Experimental): Treatment-naive AIH patients consenting to participate. This group will receive Cyclosporine-A according to a set protocol.
  Interventions: Drug: Cyclosporine-A

INTERVENTIONS:
Drug: Cyclosporine-A — Cyclosprorine-A will be administered to patients in group-B according to a set protocol and the patients will be followed at regular intervals with appropriate checking of clinical and para-clinical data.

SUMMARY:
Untreated Autoimmune hepatitis (AIH) is a progressive disease. Mainstay of treatment are corticosteroids (CS). In addition to being ineffective a substantial minority of cases, corticosteroid side-effects hamper effective therapy in another subgroup. Alternative options for induction of remission are limited. There are reports of successful salvage therapy with Cyclosporine-A (CsA) in steroid refractory cases. In addition, open-labeled studies have shown efficacy of Cyclosporine-A in treatment-naive AIH patients. There are no studies comparing CsA and CS in a head to head trial. The investigators aim to assess the efficacy and tolerability of CsA directly to the CS for induction of remission in treatment-naive AIH patients.

ELIGIBILITY:
Inclusion Criteria:

* 16-65 years old individuals with probable of definite AIH according to the revised AIH criteria.
* Willing and able to participate in the study

Exclusion Criteria:

* Non-consenting patients
* decompensated cirrhosis, i.e. clinical ascites, hepatic encephalopathy, history of variceal bleeding
* Presence of serious concomitant cardiovascular, pulmonary or renal condition
* Presence of active malignant disorder

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-12; Primary Completion 2013-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Remission | 12 months
  AST/ALT less than 2x UNL No clinical symptom
Treatment failure | 3 months
  Failure to achieve AST/ALT less than 2x UNL despite adjusting dose according to protocol

SECONDARY OUTCOMES:
Frequency of adverse events | 12 months
  Any adverse event (related or unrelated to the study drug) occuring during the induction phase.
Serious adverse event | 12 months
  Any adverse event requiring hospitalization or leading to disability or death

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Disease Research Center, Shariati Hospital, Tehran, Iran